CLINICAL TRIAL: NCT00470899
Title: Effect of Placental Drainage of Fetal Blood at Cesarean Section on the Incidence of Feto-Maternal Transfusion: A Randomized Controlled Trial
Brief Title: Effect of Placental Drainage of Fetal Blood at Cesarean Section on the Incidence of Feto-Maternal Transfusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lester E. Cox Medical Centers (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CH20041201
Record Dates: First submitted 2007-05-04; First posted 2007-05-08 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-05

CONDITIONS: Fetomaternal Transfusion
Keywords: Feto-maternal transfusion; Kleihauer-Betke
MeSH Terms: conditions — Fetomaternal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placental drainage (Experimental)
  Interventions: Procedure: drainage of placenta of fetal blood
- no drainage of fetal blood (No Intervention)

INTERVENTIONS:
Procedure: drainage of placenta of fetal blood
  Arms: placental drainage

SUMMARY:
Study hypothesis: umbilical cord drainage of fetal blood after delivery of the infant would reduce the incidence of feto-maternal transfusion. Patients were randomized to placental drainage or no drainage at the time of cesarean section. The incidence of fetal to maternal transfusion was noted postoperatively.

DETAILED DESCRIPTION:
86 patients were randomized to placental drainage vs. no drainage of fetal blood at the time of cesarean section. Kleihauer-Betke testing was performed within 12 hours postoperatively to assess the incidence of feto-maternal transfusion. A significant difference was found between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing cesarean section

Exclusion Criteria:

* Preoperative Kleihauer-Betke, known antepartum erythrocyte sensitization, overt vaginal bleeding, history of a previous delivery by low vertical cesarean section, prolonged rupture of membranes, twin gestation, failure to obtain both preoperative and postoperative Kleihauer-Betke tests.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-01; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Presence/absence of fetal blood in maternal circulation | within 12 hours postoperatively

SECONDARY OUTCOMES:
no secondary outcome measures | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Laird A Bell, MD, MPH, Study Director — Lester E. Cox Medical Center

REFERENCES:
- [Derived] Leavitt BG, Huff DL, Bell LA, Thurnau GR. Placental drainage of fetal blood at cesarean delivery and feto maternal transfusion: a randomized controlled trial. Obstet Gynecol. 2007 Sep;110(3):608-11. doi: 10.1097/01.AOG.0000277262.80793.0d. PMID 17766607